CLINICAL TRIAL: NCT03694925
Title: Diagnostic Utility of a Novel Point-of-Care Test of Calprotectin for Revision Total
Brief Title: Diagnostic Utility of a Novel Point-of-Care Test of Calprotectin for Revision Total Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Carlos Higuera-Rueda, Chairman, The Cleveland Clinic
Other Study IDs: 18-882
Record Dates: First submitted 2018-10-02; First posted 2018-10-03 (Actual); Results first posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-11

CONDITIONS: Prosthetic Joint Infection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Primary total knee arthroplasty: Primary TKA patients included in the study, to provide a baseline level for calprotectin.
  Interventions: Diagnostic Test: Calprotectin test
- Aseptic revision total knee arthroplasty: Aseptic revision TKA patients included in the study. These are patients who are not considered infected according to Musculoskeletal Infection Society criteria for infection.
  Interventions: Diagnostic Test: Calprotectin test
- Revision septic total knee arthroplasty: Septic revision TKA patients included in the study. These are patients who are considered infected according to Musculoskeletal Infection Society criteria for infection.
  Interventions: Diagnostic Test: Calprotectin test

INTERVENTIONS:
Diagnostic Test: Calprotectin test — Calprotectin will be measured both by ELISA and point of care test.

SUMMARY:
The purpose of this study is to investigate whether there are quantifiable differences in the level of calprotectin in the synovial fluid that allow separation of different modes of joint implant failure (e.g. infected, aseptic loosening). A subset of primary TKA patients (with history of OA) will be included as a baseline.

DETAILED DESCRIPTION:
Calprotectin is a biomarker closely associated with leucocytes in general, and is present in high volumes in neutrophil cells. Calprotectin is also produced by infiltrating monocytes and macrophages, where calprotectin is released upon phagocytosis. In neutrophils, calprotectin is stored intracellularly and are released upon activation of the cell. The determination of number of neutrophils and proportion of neutrophils out of total number of inflammatory cells is a diagnostic strategy commonly used in diagnosis of infection. Upon encounter with a pathogen, neutrophils have several strategies to fight infections , and produce high-levels of calprotectin. Activation of neutrophils, and release of calprotectin, can be for any reason causing activation of the complement system and aseptic Inflammatory responses. Moreover, Calprotectin is a danger associated molecular patterns (DAMP) signal influencing the inflammatory responses. The level of activated neutrophils in PJI provide basis of the presence of calprotectin in the synovial fluid of PJI patients, and thus, for calprotectin as a potential biomarker for PJI. Calprotectin-levels in the synovial fluid do not merely reflect the level of leucocytes and neutrophils present in the synovial fluid, but levels are correlated to the WBC content. Calprotectin is likely to reflect the number of activated cells and surpass the diagnostic accuracy of total WBC counts and neutrophil percentage for PJI diagnosis.

A level of calprotectin of 50 mg/L in the synovial fluid has very good diagnostic accuracy for PJI, supported by area under the curve values of more than 0.9. In a subgroup analysis for patients with chronic PJI, a NPV of 97% was observed. The excellent NPV may assist in the orthopaedic clinic to rule out the presence of infection and consider diagnostic alternatives for aseptic loosening and pain revision of the joint patient. A rapid and accurate distinction between these two causes is important as PJI and aseptic loosening are managed differently with regards to surgical Intervention and followup.

Point of Care Test diagnostics by lateral flow devices provides reliable test results within minutes of sample collection. Currently, Calprotectin can be detected by such lateral flow devices (developed by Orthogenics, Tromsø, Norway). The speed and ease of use of this test allows for diagnosis at patient's bed side. These tests can be applied in the physician's office, operating room, an ambulance, the home, the field, or in the hospital. As the results are timely they allow rapid diagnostic and identifies treatment alternatives for the patient. This technology empowers clinicians to make decisions at the "point-of-care" and can have significant impact on health care delivery and ability to address challenges of health disparities. However, it is important to validate the diagnostic utility of calprotectin POC in a diverse set of patients undergoing revision arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥18 years of age
* Patient with a diagnosis of OA (for primary TKA only)
* Subject has had no recent injections or surgeries of the joint (within past 6 weeks)
* Subject has or will have all of the medical tests required to allow MSIS classification
* Subject signs informed consent form

Exclusion Criteria:

* Subjects with a diagnostic synovial fluid specimen collection within the past 7 days
* Results are not available for medical tests required to perform MSIS classification
* Sample was obtained via lavage
* Quantity not sufficient (at least 1 ml required)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Three groups:
  Primary total knee arthroplasty Aseptic revision total knee arthroplasty Septic revision total knee arthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2020-01-07 (Actual); Study Completion 2020-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Higuera, MD, Principal Investigator — The Cleveland Clinic
Locations (2):
- United States (2):
  - Cleveland Clinic Florida, Weston, Florida
  - Cleveland Clinic, Cleveland, Ohio

IPD SHARING:
Plan to Share IPD: No
The only group we will be sharing data with is the company (Lyfstone) which is funding the research.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Primary Total Knee Arthroplasty | Aseptic Revision Total Knee Arthroplasty | Revision Septic Total Knee Arthroplasty
Started | 30 | 73 | 53
Completed | 30 | 70 | 53
Not Completed | 0 | 3 | 0
Not completed — Inadequate laboratory testing | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Primary Total Knee Arthroplasty | Aseptic Revision Total Knee Arthroplasty | Revision Septic Total Knee Arthroplasty | Total
Number analyzed (Participants) | 30 | 70 | 53 | 153
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.2 (9.8) | 65.4 (10.6) | 68.8 (10.2) | 66.9 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 40 | 26 | 83
  Male | 13 | 30 | 27 | 70
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 11 | 6 | 22
  White | 25 | 58 | 47 | 130
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 34.2 (5.9) | 32.0 (6.2) | 34.2 (9.7) | 33.2 (7.6)
Charlson Comorbidity Index [Mean (Standard Deviation); unit: units on a scale from 0 to 27] — The Charlson Comorbidity Index is a method of categorizing comorbidities of patients based on the International Classification of Diseases (ICD) diagnosis codes found in administrative data, such as hospital abstracts data. Each comorbidity category has an associated weight (from 1 to 6), based on the adjusted risk of mortality or resource use, and the sum of all the weights results in a single comorbidity score for a patient. Points are additionally added for age based on decade of life. A score of zero indicates that no comorbidities were found. Minimum is 0. Max is 27.
  units on a scale from 0 to 27 | 3.4 (2.0) | 3.4 (1.9) | 4.6 (2.5) | 3.8 (2.2)
Erythrocyte Sedimentation Rate [Mean (Standard Deviation); unit: mm/hr] — An erythrocyte sedimentation rate (ESR) is a type of blood test that measures how quickly erythrocytes (red blood cells) settle at the bottom of a test tube that contains a blood sample. Normally, red blood cells settle relatively slowly. A faster-than-normal rate may indicate inflammation in the body. Population: ESR was not collected for primary TKA as it is not standard of care ESR was not ordered by the physician for 2 septic cases
  mm/hr
    number analyzed (Participants) | 0 | 70 | 51 | 121
    (all) |  | 14 (11) | 57 (35) | 33 (32)
C Reactive Protein [Mean (Standard Deviation); unit: mg/dl] — C-reactive protein (CRP) is a protein made by the liver. CRP levels in the blood increase when there is a condition causing inflammation somewhere in the body. A CRP test measures the amount of CRP in the blood to detect inflammation due to acute conditions or to monitor the severity of disease in chronic conditions. Population: CRP was not collected for primary TKA as it is not standard of care CRP was not ordered by the physician for the 1 septic case
  mg/dl
    number analyzed (Participants) | 0 | 70 | 52 | 122
    (all) |  | 0.6 (0.7) | 11.8 (14.6) | 5.4 (11.0)
Synovial WBC Count [Mean (Standard Deviation); unit: cells/ micro liter] — Population: Synovial WBC was not collected for primary TKA as it is not standard of care Synovial WBC was unable to be run due to insufficient quantity for the 1 septic case
  cells/ micro liter
    number analyzed (Participants) | 0 | 70 | 52 | 122
    (all) |  | 735 (856) | 57803 (66595) | 25059 (51598)
Synovial PMN% [Mean (Standard Deviation); unit: percentage of cells] — Population: Synovial PMN% was not collected for primary TKA as it is not standard of care Synovial PMN% was unable to be run due to insufficient quantity for 2 septic cases
  percentage of cells
    number analyzed (Participants) | 0 | 70 | 51 | 121
    (all) |  | 21 (24) | 89 (13) | 50 (39)
Current Smoker [Count of Participants; unit: Participants] | 1 | 5 | 7 | 13
Type of Surgery [Count of Participants; unit: Participants]
  Aseptic Revision | 0 | 68 | 0 | 68
  DAIR | 0 | 1 | 18 | 19
  1st Stage of a 2 Stage | 0 | 1 | 34 | 35
  1 Stage | 0 | 0 | 1 | 1
  Primary | 30 | 0 | 0 | 30
Calprotectin POC Result [Count of Participants; unit: Participants] — Low Risk is defined 0-14 mg/L Medium Risk is defined as 14-50 mg/L High Risk is defined as >50 mg/L
  The risk refers to risk of PJI
  Participants
    Low Risk | 29 | 61 | 1 | 91
    Moderate Risk | 0 | 6 | 0 | 6
    High Risk | 1 | 3 | 52 | 56
Calprotectin ELISA Result [Count of Participants; unit: Participants] — Low Risk is defined 0-14 mg/L Medium Risk is defined as 14-50 mg/L High Risk is defined as >50 mg/L
  The risk refers to risk of PJI
  Participants
    Low Risk | 29 | 58 | 1 | 88
    Moderate Risk | 0 | 9 | 0 | 9
    High Risk | 1 | 3 | 52 | 56
Sinus Tract [Count of Participants; unit: Participants] — A tunneling wound or sinus tract is a narrow opening or passageway extending from a wound underneath the skin in any direction through soft tissue and results in dead space with potential for abscess formation.
  This was observed during surgery and collected from the operative note. This is not an outcome measure, rather it is used to assist in classifying a case as septic or aseptic using the Musculoskeletal Infection Society criteria for PJI. By definition all patients with a sinus tract are septic, however not all septic cases have a sinus tract. Population: MSIS criteria was only applied to septic and aseptic cases.
  Participants
    number analyzed (Participants) | 0 | 70 | 53 | 123
    (all) | 0 | 0 | 14 | 14
Cultures [Count of Participants; unit: Participants] — Population: Cultures were not ordered on primary TKAs as they are not standard of care
  Participants
    2 or more positive cultures: number analyzed (Participants) | 0 | 70 | 53 | 123
    2 or more positive cultures |  | 0 | 33 | 33
    1 positive culture: number analyzed (Participants) | 0 | 70 | 53 | 123
    1 positive culture |  | 9 | 47 | 56
    0 positive cultures: number analyzed (Participants) | 0 | 70 | 53 | 123
    0 positive cultures |  | 62 | 6 | 68
Histopathology [Count of Participants; unit: Participants] — Population: Histopathology was not ordered on primary TKAs as they are not standard of care.
  It was not ordered for a number septic and aseptic cases due to the individual preferences of the surgeon.
  Participants
    Positive: number analyzed (Participants) | 0 | 66 | 38 | 104
    Positive |  | 3 | 33 | 36
    Negative: number analyzed (Participants) | 0 | 66 | 38 | 104
    Negative |  | 63 | 5 | 68

OUTCOME MEASURES:

1. Primary Outcome: Calprotectin POC
Description: lateral flow point of care test
Time Frame: Day of surgery
Measure: Count of Participants; unit: Participants
Groups:
- Primary Total Knee Arthroplasty: There will be n=30 primary TKA patients included in the study, to provide a baseline level for calprotectin.
  Calprotectin test: Calprotectin will be measured both by ELISA and point of care test.
- Aseptic Revision Total Knee Arthroplasty: There will be n=70 aseptic revision TKA patients included in the study. These are patients who are not considered infected according to Musculoskeletal Infection Society criteria for infection.
  Calprotectin test: Calprotectin will be measured both by ELISA and point of care test.
- Revision Septic Total Knee Arthroplasty: There will be n=50 septic revision TKA patients included in the study. These are patients who are considered infected according to Musculoskeletal Infection Society criteria for infection.
  Calprotectin test: Calprotectin will be measured both by ELISA and point of care test.
Arm/Group | Primary Total Knee Arthroplasty | Aseptic Revision Total Knee Arthroplasty | Revision Septic Total Knee Arthroplasty
Number analyzed (Participants) | 30 | 70 | 53
Participants
  Positive at >50 mg/L | 1 | 3 | 52
  Negative at >50 mg/L | 29 | 67 | 1
  Positive at >14 mg/L | 1 | 9 | 52
  Negative at >14 mg/L | 29 | 61 | 1
Statistical Analysis 1: Comparison: Aseptic Revision Total Knee Arthroplasty vs Revision Septic Total Knee Arthroplasty; Test type: Other; Specificity = .871 — Specificity was calculated using 2x2 tables using >14 mg/L cut off. The numerator is the number of the true negatives and the denominator is the number of total negatives
Statistical Analysis 2: Comparison: Aseptic Revision Total Knee Arthroplasty vs Revision Septic Total Knee Arthroplasty; Test type: Other; Specificity = .957 — Specificity was calculated using 2x2 tables using >50 mg/L cut off. The numerator is the number of the true negatives and the denominator is the number of total negatives
Statistical Analysis 3: Comparison: Aseptic Revision Total Knee Arthroplasty vs Revision Septic Total Knee Arthroplasty; Test type: Other; Sensitivity = .981 — Sensitivity was calculated using 2x2 tables using >14 mg/L cut off. Sensitivity is the number of true positives over the number of total positives
Statistical Analysis 4: Comparison: Aseptic Revision Total Knee Arthroplasty vs Revision Septic Total Knee Arthroplasty; Test type: Other; Sensitivity = .981 — Sensitivity was calculated using 2x2 tables using >50 mg/L cut off. Sensitivity is the number of true positives over the number of total positives
Statistical Analysis 5: Comparison: Aseptic Revision Total Knee Arthroplasty vs Revision Septic Total Knee Arthroplasty; Test type: Other; Positive predictive value = .852 — Positive predictive value was calculated using 2x2 tables using >14 mg/L cut off. The numerator is the septic positives and the denominator are the total positives
Statistical Analysis 6: Comparison: Aseptic Revision Total Knee Arthroplasty vs Revision Septic Total Knee Arthroplasty; Test type: Other; Positive predictive value = .945 — Positive predictive value was calculated using 2x2 tables using >50mg/L cut off. The numerator is the septic positives and the denominator are the total positives
Statistical Analysis 7: Comparison: Aseptic Revision Total Knee Arthroplasty vs Revision Septic Total Knee Arthroplasty; Test type: Other; Negative predictive value = .984 — Negative predictive value was calculated using 2x2 tables using >14 mg/L cut off. The numerator is the aseptic negatives and the denominator is the number of total negatives
Statistical Analysis 8: Comparison: Aseptic Revision Total Knee Arthroplasty vs Revision Septic Total Knee Arthroplasty; Test type: Other; Negative predictive value = .985 — Negative predictive value was calculated using 2x2 tables using >50 mg/L cut off. The numerator is the aseptic negatives and the denominator is the number of total negatives

2. Secondary Outcome: Calprotectin ELISA
Description: ELISA analysis
Time Frame: Day of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Primary Total Knee Arthroplasty | Aseptic Revision Total Knee Arthroplasty | Revision Septic Total Knee Arthroplasty
Number analyzed (Participants) | 30 | 70 | 53
Participants
  Positive at >50 mg/L | 1 | 3 | 52
  Negative at >50 mg/L | 29 | 67 | 1
  Positive at >14 mg/L | 1 | 12 | 52
  Negative at >14 mg/L | 29 | 58 | 1
Statistical Analysis 1: Comparison: Aseptic Revision Total Knee Arthroplasty vs Revision Septic Total Knee Arthroplasty; Test type: Other; Specificity = .829 — Specificity was calculated using 2x2 tables using >14 mg/L cut off. The numerator is the number of the number of aseptic negatives and the denominator is the number of aseptics
Statistical Analysis 2: Comparison: Aseptic Revision Total Knee Arthroplasty; Test type: Other; Specificity = .957 — Specificity was calculated using 2x2 tables using >50 mg/L cut off. The numerator is the number of the number of aseptic negatives and the denominator is the number of aseptics
Statistical Analysis 3: Comparison: Aseptic Revision Total Knee Arthroplasty vs Revision Septic Total Knee Arthroplasty; Test type: Other; Sensitivity = .981 — Sensitivity was calculated using 2x2 tables using >14 mg/L cut off. Sensitivity is the number of septic positives over the number of septics
Statistical Analysis 4: Comparison: Aseptic Revision Total Knee Arthroplasty vs Revision Septic Total Knee Arthroplasty; Test type: Other; Sensitivity = .981 — Sensitivity was calculated using 2x2 tables using >50 mg/L cut off. Sensitivity is the number of septic positives over the number of septics
Statistical Analysis 5: Comparison: Aseptic Revision Total Knee Arthroplasty vs Revision Septic Total Knee Arthroplasty; Test type: Other; Positive predictive value = .813 — [estimate comment as in outcome 1, analysis 5]
Statistical Analysis 6: Comparison: Aseptic Revision Total Knee Arthroplasty vs Revision Septic Total Knee Arthroplasty; Test type: Other; Positive predictive value = .945 — [estimate comment as in outcome 1, analysis 6]
Statistical Analysis 7: Comparison: Aseptic Revision Total Knee Arthroplasty vs Revision Septic Total Knee Arthroplasty; Test type: Other; Negative predictive value = .983 — [estimate comment as in outcome 1, analysis 7]
Statistical Analysis 8: Comparison: Aseptic Revision Total Knee Arthroplasty vs Revision Septic Total Knee Arthroplasty; Test type: Other; Negative predictive value = .985 — [estimate comment as in outcome 1, analysis 8]; Negative predictive value was calculated using 2x2 tables using >50 mg/L cut off. NPV=98.5%

3. Post Hoc Outcome: Area Under the Curve
Description: Area under the curve (AUC) was calculated using receiver operator characteristic (ROC) curve using the two cut offs (>14 mg/L and >50 mg/L) for both the ELISA and POC tests. Data were collected intraoperatively during the patient's arthroplasty surgery.
  AUC - ROC curve is a performance measurement for classification problem at various thresholds settings. ROC is a probability curve and AUC represents degree or measure of separability. It tells how much model is capable of distinguishing between classes. Higher the AUC, better the model is at predicting 0s as 0s (aseptics that are negative) and 1s as 1s (septics that are positive). 1.000 represents accurately predicting each aseptic as negatve and each septic as positive. While a 0.000 represents accurately predicting each aseptic as positive and each septic as negative.
Time Frame: From completion of first patient's ELISA and POC test to last patient's ELISA and POC test
Population: Primary TKAs were no analyzed as AUC is a binary analysis representing the accuracy of predicting the correct diagnosis, ie (an aseptic is an negative, or a septic is positive). Arms/Groups are combined as the data represents the accuracy of all septics and aseptics combined at a given threshold for either the POC or ELISA test. This assessment was pre-specified to combine Arms.
Measure: Number (95% Confidence Interval); unit: probability
Groups:
- Combined Revision Total Knee Arthroplasty: All revision TKA patients included in the study.
  Calprotectin test: Calprotectin will be measured both by ELISA and point of care test.
Arm/Group | Primary Total Knee Arthroplasty | Combined Revision Total Knee Arthroplasty
Number analyzed (Participants) | 0 | 123
probability
  POC Test >50 mg/L |  | 0.969 [0.934 to 1.000]
  POC Test >14 mg/L |  | 0.926 [0.875 to 0.978]
  ELISA Test >50 mg/L |  | 0.969 [0.934 to 1.000]
  ELISA Test >14 mg/L |  | 0.905 [0.847 to 0.962]

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the the collection of the synovial fluid sample on the day of surgery which was approximately 10 minutes from incision
Description: The clinicaltrials.gov definition was used
Arm/Group | Primary Total Knee Arthroplasty | Aseptic Revision Total Knee Arthroplasty | Revision Septic Total Knee Arthroplasty
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/73 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/73 | 0/53
Other Adverse Events (participants affected / at risk) | 0/30 | 0/73 | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-17): https://cdn.clinicaltrials.gov/large-docs/25/NCT03694925/Prot_SAP_000.pdf